CLINICAL TRIAL: NCT07085728
Title: A Randomized Phase II Trial Comparing Daratumumab-Bortezomib-Dexamethasone Versus Cyclophosphamide-Bortezomib-Dexamethasone in Newly Diagnosed Multiple Myeloma With Light Chain Cast Nephropathy (LCCN)
Brief Title: Testing the Investigational Agent Combination of Daratumumab, Bortezomib, and Dexamethasone Compared to the Usual Treatment of Cyclophosphamide, Bortezomib, and Dexamethasone in Newly Diagnosed Multiple Myeloma Patients With Kidney Failure
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Eastern Cooperative Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EAA241
Record Dates: First submitted 2025-06-27; First posted 2025-07-25 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Myeloma Multiple
Keywords: EAA241; LCCN; Light Chain Cast Nephropathy; Newly Diagnosed; Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Cyclophosphamide; Injections; Bortezomib; Drugs, Generic; Dexamethasone; Calcium Dobesilate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ARM A (Cy-Bor-Dex) (Active Comparator): Cyclophosphamide-Bortezomib-Dexamethasone (4 cycles)
  Interventions: Drug: Cyclophosphamide; Drug: Bortezomib (VELCADE); Drug: Dexamethasone
- ARM B (Dara-Bor-Dex) (Experimental): Daratumumab-Bortezomib-Dexamethasone
  Interventions: Drug: Bortezomib (VELCADE); Drug: Dexamethasone; Drug: Daratumumab-hyaluronidase

INTERVENTIONS:
Drug: Cyclophosphamide — Arm A
  Other Names: Cytoxan; cyclophosphamide for injection
  Arms: ARM A (Cy-Bor-Dex)
Drug: Bortezomib (VELCADE) — Arm A, Arm B
  Other Names: bortezomib injection (generic); Velcade
Drug: Dexamethasone — Arm A, Arm B
  Other Names: Decadron
Drug: Daratumumab-hyaluronidase — Arm B
  Other Names: Darzalex FASPRO®
  Arms: ARM B (Dara-Bor-Dex)

SUMMARY:
This study is being done to answer the following question:

Can the addition of daratumumab-hyaluronidase to the usual treatment of bortezomib and dexamethasone improve kidney function in patients who are newly diagnosed with multiple myeloma and have kidney failure? This study is being done because the investigators want to find out if this approach is better or worse than the usual approach for the participant's newly diagnosed multiple myeloma. The usual approach is defined as care most people get for multiple myeloma.

If the participant decides to take part in this study, they will either get the study medications daratumumab-hyaluronidase, bortezomib, and dexamethasone for four months (4 cycles), or the typical medications used to treat your cancer (cyclophosphamide, bortezomib, and dexamethasone) for 4 months (4 cycles).

After the participant finishes their study treatment, their doctor will continue to follow their condition for 10 years to watch them for side effects and monitor their disease status. Their doctor will follow up with them every 3 months for years 1 and 2 and then every 6 months for years 3 through 10.

DETAILED DESCRIPTION:
2.1 Primary Objectives 2.1.1 To determine whether incorporation of daratumumab-hyaluronidase into the treatment algorithm for newly diagnosed light chain cast nephropathy (LCCN) will improve efficacy measured by renal response rates (RRR) per International Myeloma Working Group (IMWG) renal response criteria over 4 cycles of treatment.

2.2 Secondary Objectives 2.2.1 To evaluate the safety profile of daratumumab-hyaluronidase replacing cyclophosphamide in combination with bortezomib and dexamethasone and to compare treatment-related grades 3-5 adverse event rates based on CTCAE criteria 2.2.2 To evaluate the myeloma response per IMWG uniform response criteria over 4 cycles of therapy 2.2.3 To evaluate progression-free and overall survival

2.3 Exploratory Objectives 2.3.1 To characterize renal function over time 2.3.2 To assess stem cell mobilization initiation and collection yield in patients eligible for autologous stem cell transplant (ASCT) who undergo mobilization 2.3.3 To assess rate of eligible patients undergoing ASCT 2.3.4 To assess treatment exposure and adherence 2.3.5 To assess the association of renal impairment stage at baseline and renal response with survival outcomes

ELIGIBILITY:
3.1.1 Patient must be ≥ 18 years of age. 3.1.2 Patient must have an ECOG Performance Status 0-2. NOTE: ECOG Performance Status 3 patients are eligible if attributable to pathological fractures and/or cancer-related bone pain.

3.1.3 Patient must have multiple myeloma and meet BOTH of the following criteria for the original diagnosis of myeloma following the International Myeloma Working Group (IMWG) myeloma diagnostic criteria within 90 days prior to randomization.

1. Bone marrow plasmacytosis with ≥ 10% plasma cells or sheets of plasma cells or biopsy proven plasmacytoma.

   Plasma cell % on Bone Marrow ______ (%) Date of test:_______ Tissue biopsy of any bone lesion or extramedullary plasmacytoma if applicable (Positive / Negative for Clonal Plasma Cells) Date of test:_______
2. Any one or more of the following myeloma-defining events:

   * Anemia (hemoglobin value of >2 g/dL below the lower limit of normal, or a hemoglobin value <10 g/dL)
   * Hypercalcemia (serum calcium >1 mg/dL higher than the upper limit of normal or >11 mg/dL)
   * Bone disease (one or more osteolytic lesions on skeletal radiography, CT, or FDG-PET/CT)
   * Renal dysfunction (creatinine clearance < 40 mL/min or serum creatinine >2 mg/dL).
   * Clonal BMPCs ≥60%
   * Involved: uninvolved serum free light chain ratio ≥100
   * > 1 focal lesions on MRI studies ≥5 mm NOTE: Patients with smoldering myeloma (serum m protein ≥ 3 gm/dL or bone marrow plasma cells ≥ 10% plus no evidence of anemia, hypercalcemia, lytic bone lesions or renal dysfunction) and monoclonal gammopathy of undetermined significance (serum m protein < 3 gm/dL and bone marrow plasma cells < 10% plus no evidence of anemia, hypercalcemia, lytic bone lesions or renal dysfunction) are not eligible.

3.1.4 Patient must have newly diagnosed (within the last 90 days) light chain cast nephropathy (LCCN) defined as patients with >1 g/dl proteinuria with <10% albuminuria, and/or an involved serum free light chain (FLC) concentration >150 mg/dL.

3.1.5 Patient must have new onset of renal failure (within the last 90 days). Patient must have met one of the following criteria:

* Any serum creatinine who have an eGFR of <40 ml/min/1.73 m2 calculated with the Modification of Diet in Renal Disease (MDRD) formula
* Serum creatinine >2 mg/dL
* On dialysis NOTE: eGFR must be < 50 ml/min/1.73 m2 if eligible based on serum creatinine level and/or dialysis.

NOTE: The MDRD formula38 (mL/min/1.73 m2) = GFR = 175 x SCr-1.154 × age-0.203 × 0.742 (if female) × 1.212 (if black) SCr: ________ Date of Test: _____________ GFR: _____ (mL/min/1.73 m2) Date of calculation: ________ 3.1.6 Patient may have received myeloma targeting therapy including any of the following: cyclophosphamide, bortezomib and/or dexamethasone, as long as it was no more than one cycle AND the last dose administered was within 30 days prior to randomization.

NOTE: There is no washout period required. 3.1.7 Patient may have received plasma exchange to treat LCCN within 30 days prior to randomization.

3.1.8 Patient must not have been exposed to any prior or currently be on any anti-CD38 monoclonal antibodies.

3.1.9 Patients who have received prior investigational drug (including investigational vaccine) or invasive investigational medical device for any indication must have recovered from clinically significant adverse events prior to randomization.

3.1.10 Patient must not have current or prior exposure to focal radiation therapy within 14 days prior to randomization with the exception of palliative radiotherapy for symptomatic management but not on measurable extramedullary plasmacytoma.

3.1.11 Patient must have SPEP, UPEP, and serum FLC assays performed within 28 days prior to randomization. In addition, a bone marrow biopsy and/or aspirate and/or tissue biopsy of any bone lesion or extramedullary plasmacytoma is required to be performed within 28 days prior to randomization.

Serum M-protein by SPEP: _______ (g/dL) Date of SPEP test:_______ Urine M-protein by 24 hr UPEP: _______ (mg/24 hr) Date of UPEP test:_______ NOTE: UPEP (on a 24 hour collection) is required, no substitute method is acceptable. Urine must be followed monthly if the baseline urine M-spike is ≥ 200 mg/24 hr. If both serum and urine M-components are measurable, both must be followed in order to confirm response.

Serum Free Light Chain Assay Date of Light Chain Assay test:_______ Kappa FLC:_______ (mg/dL) or _______ (mg/L) Lambda FLC:_______ (mg/dL) or _______ (mg/L) Kappa/lambda ratio:_______ NOTE: The serum free light chain test is required to be done monthly if the patient does not have measurable disease in the serum or urine.

3.1.12 Patient must have adequate bone marrow function as defined below (these labs must be obtained < 28 days prior to randomization): Hemoglobin ≥ 7.5 g/dL (≥ 4.65 mmol/L). Use of prior red blood cell (RBC) transfusion or recombinant human erythropoietin use is permitted.

Hgb: __________ Date of Test:__________ Absolute Neutrophil Count (ANC) > 1000 mcL ANC:__________ Date of Test:__________ Platelets > 75,000 mcL. Prior platelet transfusion is permitted. Platelets:__________ Date of Test:__________ 3.1.13 Patient must have adequate hepatic function as defined below (these labs must be obtained ≤ 28 days prior to randomization): Total bilirubin ≤ 1.5 x institutional upper limit of normal (ULN) Total Bilirubin:__________ Institutional ULN:_________ Date of Test:__________ AST(SGOT) and ALT(SGPT) ≤ 3 × institutional ULN AST:_______ Institutional ULN:_________ Date of Test:_______ ALT: _______Institutional ULN:_________ Date of Test:_______ 3.1.14 Patient must not be pregnant or breast-feeding due to the potential harm to an unborn fetus and possible risk for adverse events in nursing infants with the treatment regimens being used.

All patients of childbearing potential must have a blood test or urine study within 14 days prior to randomization to rule out pregnancy.

A patient of childbearing potential is defined as anyone, regardless whether they have undergone tubal ligation, who meets the following criteria: 1) has achieved menarche at some point, 2) has not undergone a hysterectomy or bilateral oophorectomy; or 3) has not been naturally postmenopausal (amenorrhea following cancer therapy does not rule out childbearing potential) for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months).

Patient of child bearing potential? ______ (Yes or No) Date of blood test or urine study: ___________ 3.1.15 Patient must not expect to conceive or father children by using accepted and effective method(s) of contraception or by abstaining from sexual intercourse for the duration of their participation in the treatment phase of the study. Patients of childbearing potential must agree to continue contraceptive measures for at least 1 year after the last dose of Arm A protocol treatment and for at least 7 months after the last dose of Arm B protocol treatment. Patients who can father children with partners who could become pregnant must agree to continue contraceptive measures for at least 4 months after the last dose of protocol treatment. Patient must not donate eggs (ova, oocytes) or sperm while on protocol treatment and for 4 weeks after the last dose of daratumumab-hyaluronidase.

3.1.16 Patient must have the ability to understand and the willingness to sign a written informed consent document. Patients with impaired decision-making capacity (IDMC) who have a legally authorized representative (LAR) or caregiver and/or family member available will also be considered eligible.

3.1.17 Patients with a history of respiratory disease within the past 2 years (i.e. chronic obstructive pulmonary disease, moderate or severe persistent asthma) must have a forced expiratory volume in 1 second (FEV1) ≥ 50% of predicted normal (obtained within ≤ 28 days prior to randomization) to be eligible. Patients with current uncontrolled asthma of any classification are not eligible.

3.1.18 Patients with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this trial, patients should be class II or better.

3.1.19 Patients with a history of human immunodeficiency virus (HIV) must be on effective anti-retroviral therapy with an undetectable viral load within 6 months of randomization to be eligible for this trial.

3.1.20 For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated.

3.1.21 Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. Patients who completed treatment for hepatitis C at least 6 months prior to randomization and have no detectable circulating HCV are eligible.

3.1.22 Patient must not have grade 3 or 4 peripheral neuropathy at the time of randomization.

3.1.23 Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial 3.1.24 Patient must not have AL amyloidosis (amyloid light chain or primary amyloidosis), plasma cell leukemia, or CNS involvement.

3.1.25 Patient must not have known allergies, hypersensitivity, or intolerance to boron or mannitol, sorbitol, corticosteroids, monoclonal antibodies or human proteins, or their excipients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Estimated)
Dates: Start 2025-08-11 (Estimated); Primary Completion 2027-02-01 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
Renal Response Rate | Assessed every cycle on treatment up to 4 cycles (cycle duration=28 days)
  Renal response rate (RRR) is the proportion of patients achieving complete or partial renal response based on International Myeloma Working Group (IMWG) renal response criteria (Dimopoulos 2023) over 4 cycles of treatment.

SECONDARY OUTCOMES:
Grade 3-5 Overall Toxicity Rate | Assessed every cycle on treatment up to 4 cycles (cycle duration=28 days)
  Grade 3-5 overall toxicity rate is the proportion of participants who experience a maximum grade 3-5 treatment-related adverse event (AE) based on the Common Toxicity Criteria for Adverse Events Version 5.0 (CTCAEv5).
Grade 3-5 Non-Hematologic Toxicity Rate | Assessed every cycle on treatment up to 4 cycles (cycle duration=28 days)
  Grade 3-5 non-hematologic toxicity rate is the proportion of participants who experience a maximum grade 3-5 treatment-related non-hematologic AE based on CTCAEv5.
Grade 3-5 Hematologic Toxicity Rate | Assessed every cycle on treatment up to 4 cycles (cycle duration=28 days)
  Grade 3-5 hematologic toxicity rate is the proportion of participants who experience a maximum grade 3-5 treatment-related hematologic AE based on CTCAEv5.
Best Response | Assessed every cycle on treatment up to 4 cycles (cycle duration=28 days)
  Best response is the frequency of participants achieving stringent complete response (sCR), complete response (CR), partial response (PR), stable disease (SD) or disease progression (PD) based on International Myeloma Working Group (IMWG) uniform response criteria (URC; Durie 2006) over 4 cycles of treatment.
Progression-Free Survival | Disease assessed every cycle on treatment (cycle duration=28 days) and in long-term follow-up every 3 months for years 1-2 and every 6 months years 3-10
  Progression-free survival (PFS) based on the Kaplan-Meier method defined as the time from randomization until the earlier of progression (PD per IMWG URC) or death due to any cause; Patients alive without disease progression will be censored at date of last disease evaluation; Only deaths that occur within 3 months of the last disease evaluation are considered events.
Overall Survival | Assessed up to 10 years from study entry
  Overall survival (OS) based on the Kaplan-Meier method is defined as the duration of time from treatment start to date of death or censored at the date last known alive.

CONTACTS AND LOCATIONS:
Overall Officials: Amany Keruakous, Principal Investigator — ECOG-ACRIN Cancer Research Group

IPD SHARING:
Plan to Share IPD: Undecided